CLINICAL TRIAL: NCT01390519
Title: Observational Study Evaluating Efficacy, Tolerability and Treatment Algorithm of Advanced Renal Cell Cancer Patients Under Afinitor Treatment
Brief Title: A Norwegian Observational Trial Evaluating the Treatment of Advanced Renal Cell Cancer Patients Under Treatment of Afinitor
Acronym: OSAT
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CRAD001LNO03
Record Dates: First submitted 2011-06-30; First posted 2011-07-11 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Metastatic Renal Cell Carcinoma (mRCC)
Keywords: mRCC,; observational,; Afinitor,; everolimus,; 2.line
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Everolimus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — None Retained

GROUPS / COHORTS (1):
- Afinitor: Afinitor
  Interventions: Other: everolimis

INTERVENTIONS:
Other: everolimis
  Other Names: RAD001

SUMMARY:
This is a Norwegian prospective registration, observational study of patients with advanced renal cell cancer on Afinitor treatment after failure of one Tyrosine Kinase Inhibitor (TKI) ( e.g. sunitinib or sorafenib). The goal is to document the treatment algorithm of these patients in Norway and the efficacy and tolerability of Afinitor® in a pure 2.line setting.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Confirmed diagnosis of advanced renal cell cancer
* Progression on or after one VEGF -TKI (e.g. sunitibin, sorafenib)
* Written informed consent

Exclusion Criteria:

None

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced renal cell cancer whose disease has progressed on or after one VEGF-TKI therapy
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Time to progression (TTP) | maximum of 12 months after inclusion of the last patient

SECONDARY OUTCOMES:
Treatment algorithm | at end of study
  Follow up documentation
Quality of life (QoL)(EORTC-QLQ C30) | maximum of 12 months after inclusion of the last patient
  Follow up documentation
Tolerability | maximum of 12 months after inclusion of the last patient
  This will partly be assessed by registration of compliance (patient booklet), QoL and safety. Safety assessments will consist of monitoring and recording adverse events and serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- Norway (3):
  - Novartis Investigative Site, Kristiansand
  - Novartis Investigative Site, Tromsø
  - Novartis Investigative Site, Trondheim